CLINICAL TRIAL: NCT05833594
Title: Anhui Provincial Hospita
Brief Title: Whole-course Immunonutrition Combined With Chemoradiotherapy±ICIs for Local Advanced Patients With Inoperable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023WCIN001
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Immunonutrition; Inoperable
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Whole-course Immunonutrition Combined With Chemoradiotherapy±ICIs
  Interventions: Dietary Supplement: Whole-course Immunonutrition Combined With Chemoradiotherapy±ICIs
- Comparator: Whole-course nutrition Combined With Chemoradiotherapy±ICIs
  Interventions: Dietary Supplement: Whole-course Immunonutrition Combined With Chemoradiotherapy±ICIs

INTERVENTIONS:
Dietary Supplement: Whole-course Immunonutrition Combined With Chemoradiotherapy±ICIs — The Experimental group received a combination of omega-3 fatty acids, and glutamine, whereas the control group received standard formula.

SUMMARY:
Chemoradiotherapy has been a standard modality for inoperable locally advance esophageal carcinoma. The goal of this randomized control study is to compare the feasibility, and survival benefits of whole-course immunonutrition combined with chemoradiotherapy±ICIs for local advanced patients with inoperable esophageal squamous cell carcinoma. The main questions it aims to answer are: • If the feasibility and safety of whole-course immunonutrition combined with chemoradiotherapy±ICIs is better. • If the survival benefits (1, 2 and 3-years progression free survival) of whole-course immunonutrition combined with chemoradiotherapy±ICIs is longer. The Experimental group will receive a combination immunonutrition of omega-3 fatty acids, and glutamine, whereas the control group will receive standard formula.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old;
* Eastern Cooperative Oncology Group (ECOG) 0-2;
* Esophageal squamous cell carcinoma;
* cT2-4aN0-3M0 (AJCC 8th) confirmed by radiological examination;
* initial unresectable at initial diagnosis confirmed by thoracic surgeons;
* Treatment naive;
* No contraindications for adjuvant chemoradiotherapy;
* Signature of inform consent.

Exclusion Criteria:

* younger than 18 years old or older than 85 years old;
* ECOG>2;
* Esophageal adenocarcinoma, small-cell cancer and other pathological types;
* cT1anyNM0, cT4banyNM0, c anyTanyNM0 confirmed by radiological examination;
* Resectable at initial diagnosis confirmed by thoracic surgeons;
* Previous treatment of chemotherapy, radiotherapy, and other treatment;
* Contraindications for chemoradiotherapy;
* No signature of inform consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 18-85 years old;
  * Eastern Cooperative Oncology Group (ECOG) 0-2;
  * Esophageal squamous cell carcinoma;
  * cT2-4aN0-3M0 (AJCC 8th) confirmed by radiological examination;
  * initial unresectable at initial diagnosis confirmed by thoracic surgeons;
  * Treatment naive;
  * No contraindications for adjuvant chemoradiotherapy;
  * Signature of inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 1 month post treatment
  Rate of adverse events (CTCAE V4.0)
Disease Control Rate | 1 month post treatment
  Disease Control Rate

SECONDARY OUTCOMES:
1-, 2-, 3-year Progression-free survival rate (PFS). | 1 to 3 years
  1-, 2-, 3-year Progression-free survival rate (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui provincial hospital, Hefei, China

IPD SHARING:
Plan to Share IPD: Undecided